CLINICAL TRIAL: NCT03422250
Title: A Non-invasive, Multimodal Approach to Restore Functional Networks and Cognition in Alzheimer's Disease and Frontotemporal Dementia
Brief Title: Non-invasive Stimulation of Brain Networks and Cognition in Alzheimer's Disease and Frontotemporal Dementia
Acronym: NetCogBs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Michela Pievani, Principal Investigator, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GR-2011-02349787
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer's Disease; Frontotemporal Dementia, Behavioral Variant
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Alzheimer's disease (AD): anodal tDCS of the default mode network (DMN)
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Arm 2 (Experimental): Alzheimer's disease (AD): cathodal tDCS of the salience network (SN)
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Arm 3 (Experimental): Behavioral-variant frontotemporal dementia (bvFTD): anodal tDCS of the salience network (SN)
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Arm 4 (Experimental): Behavioral-variant frontotemporal dementia (bvFTD): cathodal tDCS of the default mode network (DMN)
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — 10 daily 25-minutes tDCS sessions over two weeks.

SUMMARY:
This pilot study aims to test clinical and connectivity changes following non-invasive stimulation of disease-specific networks in Alzheimer's disease (AD) and behavioral variant frontotemporal dementia (bvFTD). Brain network stimulation will be carried out with transcranial direct current stimulation (tDCS). Target networks will be the default mode network (DMN) and salience network (SN). Twenty AD and 20 bvFTD patients will be recruited and assessed with a comprehensive clinical, behavioral and cognitive battery, and 3 Tesla MRI scan (including resting-state functional MRI, arterial spin labeling, diffusion tensor imaging, structural MRI) at three time-points: baseline, after tDCS, and after 6 months. Patients will be randomized to 2 arms: anodal stimulation of the disease-specific network (DMN in AD, SN in bvFTD) or cathodal stimulation of the anti-correlated network (SN in AD, DMN in bvFTD). The intervention will consist of 10 tDCS sessions over two weeks. Cerebrospinal fluid (CSF) samples will be collected at baseline for biomarker's assessment; blood samples will be collected at each time-point to assess changes in peripheral inflammatory markers. Blood and CSF collection will be optional. A sample of 20 elderly controls will be included for baseline comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD or bvFTD according to current clinical criteria (Albert et al., 2011; Rascovsky et al., 2011)
* Ability to provide written informed consent
* Availability of a collateral source

Exclusion Criteria:

* Moderate/severe dementia
* Presence of any medical or psychiatric illness that could interfere in completing assessments

Exclusion Criteria for MRI and tDCS:

* metal implants, pace-makers, prosthetic heart valves
* claustrophobia
* history of epilepsy
* pregnancy

Exclusion Criteria for controls:

* Current or past history of clinical, neurological, or psychiatric conditions that could interfere with the assessment (e.g., transient ischemic attack, ictus, head trauma, epilepsy, multiple sclerosis, neuropathy, mood disorders, substance abuse)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2018-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michela Pievani, PhD, Principal Investigator — IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pievani M, Pini L, Cappa SF, Frisoni GB. Brain networks stimulation in dementia: insights from functional imaging. Curr Opin Neurol. 2016 Dec;29(6):756-762. doi: 10.1097/WCO.0000000000000387. PMID 27661207
- [Derived] Pini L, Pizzini FB, Boscolo-Galazzo I, Ferrari C, Galluzzi S, Cotelli M, Gobbi E, Cattaneo A, Cotelli MS, Geroldi C, Zanetti O, Corbetta M, van den Heuvel M, Frisoni GB, Manenti R, Pievani M. Brain network modulation in Alzheimer's and frontotemporal dementia with transcranial electrical stimulation. Neurobiol Aging. 2022 Mar;111:24-34. doi: 10.1016/j.neurobiolaging.2021.11.005. Epub 2021 Nov 20. PMID 34942516

RESULTS

PARTICIPANT FLOW:
Groups:
- AD: Anodal tDCS of the DMN: Alzheimer's disease (AD): anodal tDCS of the default mode network (DMN) with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: inferior parietal cortex
- AD: Cathodal tDCS of the SN: Alzheimer's disease (AD): cathodal tDCS of the salience network (SN) with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: prefrontal cortex
- bvFTD: Anodal tDCS of the SN: Behavioral-variant frontotemporal dementia (bvFTD): anodal tDCS of the salience network (SN) with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: prefrontal cortex
- bvFTD: Cathodal tDCS of the DMN: Behavioral-variant frontotemporal dementia (bvFTD): cathodal tDCS of the default mode network (DMN) with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: inferior parietal cortex
Period: Intervention
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Started | 11 | 11 | 12 | 11
Completed | 10 | 10 | 10 | 10
Not Completed | 1 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — safety (psoriasis, cortical vascular lesions on MRI) | 1 | 0 | 2 | 0
Period: Follow-up
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 8
Not Completed | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat sample (participants completing intervention)
Groups:
- AD: Anodal tDCS of the DMN: AD: anodal tDCS of the default mode (DMN) network with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: inferior parietal cortex
- AD: Cathodal tDCS of the SN: AD: cathodal tDCS of the salience network (SN) with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: prefrontal cortex
- bvFTD: Anodal tDCS of the SN: bvFTD: anodal tDCS of the salience network (SN) with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: prefrontal cortex
- bvFTD: Cathodal tDCS of the DMN: bvFTD: cathodal tDCS of the default mode network (DMN) with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: inferior parietal cortex
- Total: Total of all reporting groups
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (6) | 73 (6) | 71 (10) | 69 (11) | 71 (8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 6 | 4 | 3 | 5 | 18
  Male | 4 | 6 | 7 | 5 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 10 | 40
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Disease Severity (CDR)
Description: CDR - Clinical Dementia Rating score
  The clinical dementia rating (CDR) is a clinical global rating scale administered to both the participant and the caregiver, assessing 6 domains of participant function: memory, orientation, judgement and problem solving, community affairs, home and hobbies and personal care. Each domain is based on a 5-point scale ranging from no impairment=0, questionable impairment=0.5, mild impairment=1, moderate impairment=2 to severe impairment=3. The global CDR score is computed via a memory-weighted averaging algorithm of the six domain scores and ranges from 0 to 5. The CDR-sum of boxes (CDR-SB) is the sum of the individual domain scores and ranges from 0 to 18. Higher scores indicate more clinical impairment. Negative changes at post tDCS compared to baseline represent an improvement on the scale.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AD: Anodal tDCS of the DMN: AD: anodal tDCS of the default mode network with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: inferior parietal cortex
- AD: Cathodal tDCS of the SN: AD: cathodal tDCS of the salience network with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: prefrontal cortex
- bvFTD: Anodal tDCS of the SN: bvFTD: anodal tDCS of the salience network with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: prefrontal cortex
- bvFTD: Cathodal tDCS of the DMN: bvFTD: cathodal tDCS of the default mode network with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: inferior parietal cortex
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale
  CDR global | -0.1 (0.2) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  CDR sum of boxes | 0.1 (0.4) | 0.0 (0.2) | -0.1 (0.3) | 0.0 (0.0)

2. Primary Outcome: Change in Behavioral Symptom Severity (NPI)
Description: The Neuropsychiatric Inventory (NPI) is a behavioral scale administered to the caregiver assessing 12 dimensions: delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, euphoria, apathy, disinhibition, irritability, aberrant motor activity, nighttime behaviors, and appetite/eating. Each dimension has multiple screening questions relating to symptoms. If the answer to the screening questions is "Yes", the dimensional-score is the product of frequency (1=occasionally to 4=very frequently) and severity (1=Mild to 3=Severe) of symptoms. Dimensional-scores are summed (from 0 to 144). Higher scores indicate greater behavioral disturbances. Negative changes at post tDCS compared to baseline represent an improvement on the scale.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale | -1 (3) | -3 (6) | -1 (4) | -6 (11)

3. Primary Outcome: Change in Behavioral Symptom Severity (FBI)
Description: The Frontal Behavioral Inventory (FBI) is a 24-item inventory designed to assess behavior and personality changes via caregiver. Item-level scores range from 0=none, 1=mild/occasional, 2=moderate, 3=severe/most of the time. Item-scores are summed (from 0 to 72). Higher scores indicate greater behavioral/personality disturbances. Negative changes at post tDCS compared to baseline represent an improvement on the scale.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10
score on a scale | -2 (4) | -4 (8)

4. Primary Outcome: Change in Functional Connectivity
Description: Default mode network (DMN) and salience network (SN) mean functional connectivity is assessed on resting state functional MRI. Functional connectivity is standardized to Z scores and thresholded at Z>2. Higher values denote greater functional connectivity. A positive change at post tDCS compared to baseline represents an increase in resting-state functional connectivity.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 9 | 9
Z-score
  DMN | 0.08 (0.13) | -0.09 (0.11) | -0.02 (0.23) | -0.04 (0.15)
  SN | -0.06 (0.15) | 0.05 (0.2) | 0.08 (0.18) | 0.02 (0.12)

5. Primary Outcome: Change in Cerebral Blood Flow
Description: Default mode network (DMN) and salience network (SN) mean cerebral blood flow is assessed on arterial spin labeling. Cerebral blood flow is computed by averaging values across the DMN and SN regions of interest. Cerebral blood flow is a measure of brain perfusion, higher values denoting higher perfusion. A positive change at post tDCS compared to baseline represents an increase in perfusion.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 9 | 9 | 7 | 9
ml/100g/min
  DMN | 4.87 (8.92) | -0.06 (9.46) | 0.56 (7.72) | 3.08 (3.45)
  SN | 4.37 (7.00) | -1.92 (12.3) | 2.34 (4.84) | 1.41 (4.09)

6. Secondary Outcome: Change in Cognition: Memory
Description: The composite memory score consists of the averaged Z-standardized scores of 5 memory tests: immediate and delayed auditory verbal learning test recall, Rey-Osterrieth complex figure recall, story recall, digit span backward and forward tests. Each test score is normalized to an independent dataset of healthy controls. Z-scores have no minimum/maximum values. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values denote better memory performance. Positive changes at post tDCS compared to baseline represent an improvement in memory.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 10 | 10
z score | 0.3 (0.2) | 0.3 (0.3) | 0.1 (0.3) | 0.2 (0.3)

7. Secondary Outcome: Change in Cognition: Language
Description: The composite language score consists of the averaged Z-standardized scores of 2 language tests: verbal fluency and token tests. Each test score is normalized to an independent dataset of healthy controls. Z-scores have no minimum/maximum values. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values denote better language performance. Positive changes at post tDCS compared to baseline represent an improvement in language.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 10 | 10
z score | 0.7 (0.6) | 0.4 (0.6) | 0.7 (0.9) | 0.4 (0.6)

8. Secondary Outcome: Change in Cognition: Executive Function
Description: The composite executive function score consists of the averaged Z-standardized scores of 2 executive functions tests: trail making test part A and part B tests. Each test score is normalized to an independent dataset of healthy controls and inverted. Z-scores have no minimum/maximum values. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values denote better executive function performance. Positive changes at post tDCS compared to baseline represent an improvement in executive functions.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 10 | 10
z score | 0.3 (2.9) | -0.3 (2.4) | 0.7 (2.3) | -0.7 (1.6)

9. Secondary Outcome: Change in Cognition: Visuospatial Function
Description: The visuospatial function score consists of the Z-standardized scores for the Rey-Osterrieth complex figure copy test. Scores are normalized to an independent dataset of healthy controls. Z-scores have no minimum/maximum values. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values denote better visuospatial performance. Positive changes at post tDCS compared to baseline represent an improvement in visuospatial functions.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 10 | 10
z score | 1.2 (1.1) | 0.0 (1.6) | 0.1 (0.8) | 0.4 (0.9)

10. Secondary Outcome: Change in Cognition: Emotion Recognition
Description: The composite emotion recognition score consists of the averaged Z-standardized scores for 2 emotion recognition tests: reading the Mind in the Eyes and 60 Ekman faces tests. Each test score is normalized to an independent dataset of healthy controls. Z-scores have no minimum/maximum values. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values denote better emotion recognition performance. Positive changes at post tDCS compared to baseline represent an improvement in emotion recognition.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 10 | 10
z score | 0.1 (0.5) | 0.1 (0.6) | 0.3 (1.2) | 0.1 (0.9)

11. Secondary Outcome: Change in Structural Connectivity: FA
Description: Fractional anisotropy (FA) is assessed on diffusion weighted imaging. FA values are averaged in default mode network (DMN) and salience network (SN) regions of interest. FA values denote the directionality of water diffusivity, ranging from 0 (isotropic diffusion) to 1 (anisotropic diffusion). Higher values denote higher directionality and connectivity. Positive changes at post tDCS compared to baseline represent an improvement in the measure.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 9 | 7
score on a scale
  DMN FA | 0.000 (0.007) | -0.003 (0.006) | -0.002 (0.008) | 0.000 (0.008)
  SN FA | 0.003 (0.009) | -0.002 (0.011) | -0.002 (0.009) | 0.001 (0.011)

12. Secondary Outcome: Change in Structural Connectivity: MD, AxD, RaD
Description: Mean diffusivity (MD), axial diffusivity (AxD), and radial diffusivity (RaD) are assessed on diffusion weighted imaging. MD, AxD, RaD values are averaged in default mode network (DMN) and salience network (SN) regions of interest. MD, AxD, and RaD measure water diffusion and are expressed in mm^2/s (starting from 0 with no maximum value; scaled at x10^-3). Higher values denote higher diffusion and lower connectivity. Negative changes at post tDCS compared to baseline represent an improvement in the measure.
Time Frame: Baseline, post tDCS (week 3)
Population: Modified intention-to-treat sample (participants completing intervention)
Measure: Mean (Standard Deviation); unit: x10^-3 mm^2/s
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
Number analyzed (Participants) | 10 | 10 | 9 | 7
x10^-3 mm^2/s
  DMN MD | -0.003 (0.017) | -0.001 (0.019) | 0.007 (0.008) | 0.007 (0.008)
  SN MD | -0.004 (0.016) | -0.002 (0.017) | 0.010 (0.009) | 0.007 (0.008)
  DMN AxD | -0.004 (0.017) | -0.006 (0.024) | 0.009 (0.014) | 0.008 (0.011)
  SN AxD | -0.004 (0.017) | -0.008 (0.029) | 0.014 (0.018) | 0.010 (0.012)
  DMN RaD | -0.002 (0.017) | 0.001 (0.017) | 0.007 (0.009) | 0.006 (0.009)
  SN RaD | -0.005 (0.017) | 0.000 (0.015) | 0.008 (0.009) | 0.005 (0.011)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of enrollment to follow-up assessment (approx 6 months).
Description: A questionnaire was administered to all participants to monitor events occurring within 24 hours after each tDCS session. A questionnaire was also administered at the end of the first and last tDCS sessions to monitor the occurrence of the most common discomfort sensations related to tDCS and their intensity.
Groups:
- AD: Anodal tDCS of the DMN: AD: anodal tDCS of the default mode network (DMN) with transcranial direct current stimulation (tDCS): 10 daily 25-minutes tDCS sessions over two weeks.
  Stimulation target: inferior parietal cortex
Arm/Group | AD: Anodal tDCS of the DMN | AD: Cathodal tDCS of the SN | bvFTD: Anodal tDCS of the SN | bvFTD: Cathodal tDCS of the DMN
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 1/11
Other Adverse Events (participants affected / at risk) | 5/11 | 6/11 | 5/12 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AD: Anodal tDCS of the DMN (N=11) | AD: Cathodal tDCS of the SN (N=11) | bvFTD: Anodal tDCS of the SN (N=12) | bvFTD: Cathodal tDCS of the DMN (N=11)
Intestinal infarct (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AD: Anodal tDCS of the DMN (N=11) | AD: Cathodal tDCS of the SN (N=11) | bvFTD: Anodal tDCS of the SN (N=12) | bvFTD: Cathodal tDCS of the DMN (N=11)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 | 0
Chest pain (General disorders) | 0 | 1 (1) | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 (1) | 0 | 1 (1)
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1)
Itching (tDCS related discomfort sensation) (Skin and subcutaneous tissue disorders) | 0 | 3 (4) | 1 (1) | 1 (1)
Pain (tDCS related discomfort sensation) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0
Burning (tDCS related discomfort sensation) (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 0 | 2 (2)
Warmth/Heat (tDCS related discomfort sensation) (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0
Pinching (tDCS related discomfort sensation) (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (7) | 3 (3) | 1 (1)
Metallic/Iron taste (tDCS related discomfort sensation) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0
Fatigue (tDCS related discomfort sensations) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0
Other tDCS related discomfort sensations (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT03422250/Prot_SAP_000.pdf